CLINICAL TRIAL: NCT01629979
Title: Efficacy and Tolerance of Transplantation of Harvested Epidermal Cells and Narrow-Band UVB in Vitiligo
Brief Title: Epidermal Cell Transplantation in Vitiligo Skin
Acronym: VITICELL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-018886-52
Record Dates: First submitted 2012-03-23; First posted 2012-06-28 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: VITILIGO
MeSH Terms: conditions — Vitiligo | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Grafting of autologous epidermal harvested cells and UVB (Experimental): Grafting with epidermal cells: A superficial skin shaving excision will be obtained from pigmented skin using a dermatome. A cell suspension will be obtained by trypsinisation. Vitiligo skin will be dermabraded by Erbium: Yag laser after local anaesthesia. The cell suspension will be spread on the dermabraded skin area and fixed with dressings. Keratinocyte, and melanocyte counts will be performed on an aliquot of the cell suspension. One symmetrical patch of vitiligo will be chosen as control and left untreated.
  Narrow-band UVB treatment: Four weeks after transplantation of epidermal cells, the grafted and control patch will be treated by Narrow-band UVB. Treatment will be performed 2 times a week. Narrow-band UVB treatment will be performed for at least 3 months or 24 treatments.
  Interventions: Procedure: Grafting with epidermal cells
- UVB treatment (Active Comparator): UVB treatment twice a week during 3months
  Interventions: Radiation: UVB treatment

INTERVENTIONS:
Procedure: Grafting with epidermal cells — A superficial skin shaving excision will be obtained from pigmented skin using a dermatome. A cell suspension will be obtained by trypsinisation. Vitiligo skin will be dermabraded by Erbium: Yag laser after local anaesthesia. The cell suspension will be spread on the dermabraded skin area and fixed with dressings. Keratinocyte, and melanocyte counts will be performed on an aliquot of the cell suspension. One symmetrical patch of vitiligo will be chosen as control and left untreated.
  Narrow-band UVB treatment: Four weeks after transplantation of epidermal cells, the grafted and control patch will be treated by Narrow-band UVB. Treatment will be performed 2 times a week. Narrow-band UVB treatment will be performed for at least 3 months or 24 treatments.
  Arms: A: Grafting of autologous epidermal harvested cells and UVB
Radiation: UVB treatment — the control patch will be treated by Narrow-band UVB. Treatment will be performed 2 times a week. Narrow-band UVB treatment will be performed for at least 3 months or 24 treatments.
  Arms: UVB treatment

SUMMARY:
The effects of treatment of transplantation of harvested autologous epidermal cells on vitiligo lesions followed by narrow-band UVB will be investigated in a randomized controlled study.

DETAILED DESCRIPTION:
Introduction: Transplantation of harvested autologous epidermal cells in vitiligo is widely used in vitiligo but randomized controlled trials in the literature investigating the efficacy of these noncultured keratinocyte/melanocyte suspensions are scarce. In addition there are few data regarding the relationship between the cellular contents of epidermal suspensions and the clinical outcome.

Aim of the study: To perform a prospective, controlled, randomized, intra-individual comparative study in vitiligo lesions treated with epidermal cell transplantation with additional narrow-band UVB treatment using epidermal cell suspensions that have been characterized at the cellular level.

Study design:

Grafting with epidermal cells: A superficial skin shaving excision will be obtained from pigmented skin using a dermatome. A cell suspension will be obtained by trypsinisation. Vitiligo skin will be dermabraded by Erbium: Yag laser after local anaesthesia. The cell suspension will be spread on the dermabraded skin area and fixed with dressings. Keratinocyte, and melanocyte counts will be performed on an aliquot of the cell suspension. One symmetrical patch of vitiligo will be chosen as control and left untreated.

Narrow-band UVB treatment: Four weeks after transplantation of epidermal cells, the grafted and control patch will be treated by Narrow-band UVB. Treatment will be performed 2 times a week. Narrow-band UVB treatment will be performed for at least 3 months or 24 treatments.

Evaluation of the treatment success: The grade of pigmentation in all lesions will be evaluated clinically, with photographs. The clinical rating will be performed as follows: 0 = no repigmentation; 1 = 1-25% repigmentation; 2 = 26 to 50% repigmentation; 3 = 51 to 75% repigmentation; and 4 = 76 to 100% repigmentation. The evaluation of the photographs will be performed blinded by physicians not engaged in the treatment phase of the study. In addition the surface of vitiligo patches will be traced on transparent sheets and monitored by planimetry.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18yr
* Stable vitiligo (no lesion since 12 mo)
* 2 symmetrical vitiligo patches of at least 10 cm2
* Vitiligo requiring UVB treatment
* Women using a contraceptive

Exclusion Criteria:

* History of keloids
* History of skin cancer
* Photosensitivity
* Positive blood test for HIV, HBV, HVC, or HTLV1
* Pregnant or breastfeeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Repigmentation rate at 12 months | 12months
  Repigmentation rate at 12 months

SECONDARY OUTCOMES:
Repigmentation > 70% at 12 months | 12 months
  Repigmentation > 70% at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: philippe bahadoran, doctor, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Centre hospitalier Universitaire de Nice, Nice, France